CLINICAL TRIAL: NCT04770311
Title: Childhood Obesity Microbiome Study
Acronym: CHOICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00107438
Record Dates: First submitted 2021-02-23; First posted 2021-02-25 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Pediatric Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): In a typical Healthy Lifestyless Nutrition visit, dietitians provide medical nutrition therapy to patients and their families. This includes addressing abnormal, nutrition-related lab values and providing targeted nutrition advice (foods to include, foods to limit) in order to resolve said labs. Motivational interviewing techniques will be used to help families identify barriers to Lifestyles change and provide strategies to help overcome these barriers. Families will receive compensation per each nutritional visit.
- Intervention (Other): Besides the usual standard of care during the nutrition visits, participants will have guidance on a microbiome-friendly diet and will receive groceries 1 time per week for 4 weeks.
  Interventions: Behavioral: Microbiome friendly diet

INTERVENTIONS:
Behavioral: Microbiome friendly diet — Families in the intervention group will have a microbiome-friendly nutrition assessment and will also receive groceries one time per week for four weeks to help achieve a more microbiome-friendly diet.
  Arms: Intervention

SUMMARY:
The purpose of this study is to measure the effectiveness of a microbiome diet using direct food provision on dietary quality and microbiome composition among children with obesity. This study proposes a pilot randomized, controlled clinical trial in children of a dietary intervention informed by microbiome science.

DETAILED DESCRIPTION:
Childhood obesity is a global health crisis and contributes to shortened life expectancy in the US, with higher rates and more serious co-morbidities among minorities. Existing dietary interventions demonstrate significant heterogeneity of treatment response among diverse populations, and clear information to tailor diet to individual-level characteristics is not yet available. Recent science suggests that the gut microbiome may in part explain inter-individual variation in pediatric obesity and treatment response. Intestinal microbial communities play causal roles in models of obesity and are distinct between individuals. However, it is unknown how the microbiome mediates response to existing dietary guidelines for children with obesity.

Evidence-based nutritional standards for treatment of pediatric obesity are well-established, and aim to reduce body mass index and cardio-metabolic risk. However, these standards have not translated into reduced prevalence of obesity among children, particularly those in racially diverse and low-income groups. One explanation is the significant inter-individual variability in metabolic response to dietary interventions, suggesting that certain food components in a diet may benefit some individuals more than others. Another explanation is that dietary adherence is highly variable, and requires skills or resources not available to all people. For example, translating dietary recommendations into food procurement, preparation, and consumption requires baseline levels of educational attainment, child acceptability of foods, diet compatibility with cultural preferences, and may be seen as time-consuming. These obstacles are hard to overcome for children and families from low-income and minority groups, who are known to have low show rates and engagement in nutrition studies despite being at disproportionate risk of diseases like obesity and metabolic disease. The one-size-fits-all approach to dietary recommendations is failing the most vulnerable children in the nation.

Recent science suggests that the gut microbiome provides new opportunities to address these long-standing challenges. Microbiome transplant experiments in mice have demonstrated that increased adiposity can be conferred from bacterial communities originating from individuals with obesity. Furthermore, variation in microbiome composition between individuals can predict response to dietary intervention, suggesting a mechanism for why certain individuals lose weight on specific diets and other individuals do not. Another intriguing aspect of microbiome science is how its adoption could introduce new methodological techniques to obesity treatment. In particular, the plummeting costs and turnaround times of metagenomic DNA sequencing used in microbiome research opens new opportunities for rapidly providing biomarker information to a wide number of people. |

No evidence exists that describes microbiome signatures with objective measures of dietary quality among children with obesity. The work to be completed here will be a vital first step towards integrating the promise of microbiome science into the treatment of pediatric obesity. Our team is uniquely suited to take this step as leaders in microbiome science (David) and childhood obesity (Armstrong). By working together to predict how individual microbiome variation shapes responses to diet therapy, an important step towards personalizing dietary recommendations for children based on gut microbiome signatures that predict the best outcome will be taken. In addition, linking microbial signatures to measures of diet quality will provide researchers with much-needed molecular tools for assessing dietary compliance and intervention success. Finally, insights into the impact of receiving metagenomic data on children's' motivation towards healthy behaviors could provide behavioral and implementation scientists with new tools for improving adherence with obesity treatment

ELIGIBILITY:
Inclusion Criteria:

* Child aged 6 - 11 years (not yet aged 12)
* Child with BMI ≥ 95th percentile
* Parents are willing to accept home deliveries and have the ability to be home at the time and day that is most convenient for them to receive the groceries; or, have transportation available to go and pick up groceries at a time and date that is most convenient for them at a Walmart location.

Exclusion Criteria:

* Does the child have a current diagnosis of obesity due to an underlying condition such as hypothyroidism, Cushing's disease, or known genetic condition?
* Is the child currently taking any weight-loss medication (steroids, anti-psychotics, anti-depressants)
* Has the child started a stimulant medication in the past 3 months? (stimulants include, among others, Ritalin, Adderall, concerta, focalin, vyvanse).
* Is the child currently taking, or has taken in the past 4 weeks, an antibiotic?
* Is the child currently taking, or plans to take in the next 4 weeks, a weight loss medication?
* Is the patient on a pharmacotherapy or weight loss surgery track in Healthy Lifestyless?
* Has the patient lost more than 5% of their body weight in the preceding 6 months?

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2021-11-20 (Actual); Study Completion 2021-11-20 (Actual)

PRIMARY OUTCOMES:
Change in child dietary quality as measured by the DSQ | Baseline, week 4 and week 8
  The investigators will use the DSQ, which is the 26-item Dietary Screener Questionnaire, that asks about the frequency of consumption in the past month of selected foods and drinks. The DSQ captures intakes of fruits and vegetables, dairy/calcium, added sugars, whole grains/fiber, red meat, and processed meat. The study team will be focusing on microbiome friendly food, such as whole grains a fiber rich foods.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Armstrong, MD, Principal Investigator — Duke department of Pediatrics
Locations (1):
- Duke Healthy Lifestyles Roxboro Street, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No